CLINICAL TRIAL: NCT00470574
Title: Pilot Study of Immunization of High Risk Breast Cancer Patients With a Sialyl Lewisª -Keyhole Limpet Hemocyanin Conjugate Plus the Immunological Adjuvant QS-21
Brief Title: Vaccine Therapy and QS21 in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-156; P30CA008748 (NIH); MSKCC-06156
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — saponin QA-21V1; Immunoenzyme Techniques; Immunologic Techniques

ARMS (1):
- Vaccine Therapy and QS21 (Experimental): Patients receive sialyl Lewisª -keyhole limpet hemocyanin conjugate vaccine subcutaneously (SC) and QS21 immunoadjuvant SC once in weeks 1, 2, 3, 7, and 19 in the absence of disease progression or unacceptable disease.
  Blood samples are collected periodically and evaluated for circulating tumor cells and reactivity against sialyl Lewisª antigen in ELISA and/or immunoprecipitation-western blot assays.
  After completion of study treatment, patients are followed every 3 months
  Interventions: Biological: QS21; Biological: sialyl Lewisª-keyhole limpet hemocyanin conjugate vaccine; Other: immunoenzyme technique; Other: immunologic technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: QS21
Biological: sialyl Lewisª-keyhole limpet hemocyanin conjugate vaccine
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy together with QS21 may cause a stronger immune response and kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects and how well giving vaccine therapy together with QS21 works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of sialyl Lewisª -keyhole limpet hemocyanin conjugate vaccine and QS21 immunoadjuvant in patients with metastatic breast cancer.
* Determine the IgG and IgM antibody response to this regimen in these patients.
* Determine the proportion of breast cancer cells expressing this antigen in these patients.

Secondary

* Monitor the presence of circulating tumor cells prior to, during, and after this regimen in these patients.

OUTLINE: Patients receive sialyl Lewisª -keyhole limpet hemocyanin conjugate vaccine subcutaneously (SC) and QS21 immunoadjuvant SC once in weeks 1, 2, 3, 7, and 19 in the absence of disease progression or unacceptable disease.

Blood samples are collected periodically and evaluated for circulating tumor cells and reactivity against sialyl Lewisª antigen in ELISA and/or immunoprecipitation-western blot assays.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV breast cancer meeting 1 of the following criteria:

  * No evidence of disease
  * Stable disease on hormonal therapy

    * Stable disease must be present for ≥ 2 months and include < 30% decrease or < 20% increase in the sum of the longest diameter of target lesion
    * No new target lesions or unequivocal progression of non-target lesions
    * Elevation in the CA 153 (BR2729) or CEA values allowed
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female or male
* Menopausal status not specified
* Karnofsky performance status 80-100%
* Lymphocyte count ≥ 500/mm³
* WBC ≥ 3,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergy to seafood
* No NYHA class III-IV cardiac disease
* No other active cancers except basal cell or squamous cell carcinoma of the skin
* No active infection requiring antibiotic treatment
* No known history of immunodeficiency or autoimmune disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior surgery
* At least 6 weeks since prior immunotherapy
* No prior sialyl Lewisª antigen
* No concurrent immunosuppressive medications (i.e., corticosteroids)
* Concurrent hormonal therapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-03-20 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ann Gilewski, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine Therapy and QS21
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine Therapy and QS21
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 44 [31 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Vaccine Therapy and QS21
Number analyzed (Participants) | 0

2. Primary Outcome: Immune Response
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Vaccine Therapy and QS21
Number analyzed (Participants) | 0

3. Secondary Outcome: Presence of Circulating Tumor Cells
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Vaccine Therapy and QS21
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Vaccine Therapy and QS21
All-Cause Mortality (participants affected / at risk) | 4/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Therapy and QS21 (N=7)
Ocular/Visual - Other (specify) (Eye disorders) | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Therapy and QS21 (N=7)
Injection site reaction/extravasation (General disorders) | 7
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 3
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 3
Metabolic/Lab - Other (specify) (Metabolism and nutrition disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pain - Head/headache (Nervous system disorders) | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Edema: limb (General disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Mucositis (func/sympt)- Oral cavity (Gastrointestinal disorders) | 1
Ocular/Visual - Other (specify) (Eye disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 1
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT00470574/Prot_SAP_000.pdf